CLINICAL TRIAL: NCT03813472
Title: Validation of Skin Hydration Sensor for Atopic Dermatitis
Brief Title: Hydration Sensor for Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: SX08152018
Record Dates: First submitted 2019-01-20; First posted 2019-01-23 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Atopic Dermatitis; Healthy Children
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atopic Dermatitis: Evaluate sensor performance for hydration sensing.
  Interventions: Device: Hydration Sensor
- Healthy aged matched controls: Evaluate sensor performance for hydration sensing.
  Interventions: Device: Hydration Sensor

INTERVENTIONS:
Device: Hydration Sensor — This device includes a hydration sensor embedded within silicone and applied to the skin with a medical grade adhesive.

SUMMARY:
Pilot study of a soft, flexible hydration sensor

DETAILED DESCRIPTION:
Assessment of accuracy and feasibility of a skin hydration sensor at detecting differences in skin hydration between skin affected by atopic dermatitis and areas not affected.

ELIGIBILITY:
Inclusion Criteria:

* Children <18 years of age
* Children with new or prior atopic dermatitis diagnosis
* English speaking
* Children who are healthy, aged matched controls

Exclusion Criteria:

* Individuals who are pregnant

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Healthy, aged matched controls or children with prior diagnosis of atopic dermatitis as confirmed by clinical diagnosis by a board-certified dermatologist
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Percent Agreement | 1 hour
  Percent agreement between experimental sensor and commercially available transepidermal water loss meter.

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xu, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States